CLINICAL TRIAL: NCT04286802
Title: Impact of Self-monitoring of Salt Intake by Salt Meter in Hypertensive Patients
Acronym: SMAL-SALT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-60-21
Record Dates: First submitted 2020-02-11; First posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Hypertension; Salt; Excess
Keywords: hypertension; uncontrolled; salt, excess; salt meter
MeSH Terms: conditions — Hypertension | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salt-meter (Experimental): Patients received salt-meter in conjunction with dietary education by trained dietician to help monitoring the salt content in food, as well as usual care by their primary physicians.
  Interventions: Device: Salt-meter; Behavioral: Education
- Control (Active Comparator): Patients received dietary education by trained dietician and usual care by their primary physicians.
  Interventions: Behavioral: Education

INTERVENTIONS:
Device: Salt-meter — Salt-meter, developed by Faculty of Engineering at Mahidol University, is a device to measure sodium chloride content in the food and reflects to user with number and symbols for easy-understanding.
  Arms: Salt-meter
Behavioral: Education — Program dietary education by certified dietician who did not know the patients arm allocation.

SUMMARY:
Hypertension is one of the most common chronic medical conditions. The concerned sequelae are the cardiovascular complications, especially acute myocardial infarction and stroke. In Thailand, the incidence of hypertension is increasing each year. Many clinical studies found that salt intake over the reference level (>5 g/day) would result in elevated blood pressure (BP) and long-term morbidity. Dietary salt reduction campaigns were unsuccessful, in part, due to time limitation in the clinic, lacking of awareness, and the higher threshold to detect salt taste in chronic high salt ingestion. Salt meter is a device used to detect sodium content in daily food. It will facilitate monitoring and control of salt intake. The 24-hour urinary sodium excretion is an acceptable method to reflect the quantity of sodium intake. This study aimed to compare the efficacy of salt meter plus dietary education compared with education alone in terms of salt intake reduction, blood pressure, salt taste sensitivity, and vascular consequence.

DETAILED DESCRIPTION:
A randomized-controlled trial was conducted in hypertensive patients whose BP was uncontrolled (systolic BP ≥140 mmHg or diastolic BP ≥90 mmHg) despite therapy or antihypertensive-naïve. Patients were randomized to receive salt meter to use in conjunction with dietary education (group A) or receive education only (group B), and were followed up for 8 weeks. Dietary education was provided by certified dietician without awareness of patients' allocation. The primary endpoint was change in 24-hour urinary sodium excretion. Changes in BP, salt taste sensitivity threshold, cardio-ankle vascular index (CAVI), as well as motivation to maintain low salt diet were also analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Mean SBP 140-179 mmHg or mean DBP 90-109 mmHg (average 3 times)
* Diagnosed of hypertension for at least 3 months
* No adjustment of antihypertensive agents for at least 1 month
* 24h Urine sodium ≥ 90 mmol/day
* eGFR ≥ 45 ml/min/1.73 sq.m.

Exclusion Criteria:

* eGFR < 45 ml/min/1.73 sq.m.
* UACR > 300 mg/g
* Serum potassium > 6.0 mmol/l
* Serum sodium < 135 mmol/l
* Unable to collect 24-hour urine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-07-11 (Actual); Primary Completion 2020-02-21 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
24-hour urinary sodium excretion | 8 weeks
  Change in 24-hour urinary sodium excretion from baseline

SECONDARY OUTCOMES:
Change in systolic and diastolic blood pressure | 8 weeks
  Changes in systolic and diastolic blood pressure from baseline
Improvement in salt taste sensitivity by evaluating the salt detection or recognition thresholds | 8 weeks
  Using the different saline concentration in solution. Starting from the lowest to higher concentration, the point when the patient can differentiate from distilled water is called "detection threshold", and the point that patient can identify salty taste is called "recognition" threshold.
Change in cardio-ankle vascular index (CAVI) | 8 weeks
  Change in cardio-ankle vascular index (CAVI) from baseline

OTHER OUTCOMES:
Number of patients with hypertensive emergency | 8 weeks
  Number of patients documented to have hospitalisation for hypertension treatment including hypertensive emergency requiring intravenous antihypertensive agents.
Questionnaire about motivation to maintain low salt diet | after 8 weeks
  Scale from 0 to 10 to estimate self motivation for taking low salt strategy at baseline and at 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Ramathibodi Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mente A, O'Donnell MJ, Rangarajan S, McQueen MJ, Poirier P, Wielgosz A, Morrison H, Li W, Wang X, Di C, Mony P, Devanath A, Rosengren A, Oguz A, Zatonska K, Yusufali AH, Lopez-Jaramillo P, Avezum A, Ismail N, Lanas F, Puoane T, Diaz R, Kelishadi R, Iqbal R, Yusuf R, Chifamba J, Khatib R, Teo K, Yusuf S; PURE Investigators. Association of urinary sodium and potassium excretion with blood pressure. N Engl J Med. 2014 Aug 14;371(7):601-11. doi: 10.1056/NEJMoa1311989. PMID 25119606
- [Background] Cook NR, Kumanyika SK, Cutler JA, Whelton PK; Trials of Hypertension Prevention Collaborative Research Group. Dose-response of sodium excretion and blood pressure change among overweight, nonhypertensive adults in a 3-year dietary intervention study. J Hum Hypertens. 2005 Jan;19(1):47-54. doi: 10.1038/sj.jhh.1001775. PMID 15343354
- [Background] MacGregor GA, Markandu ND, Sagnella GA, Singer DR, Cappuccio FP. Double-blind study of three sodium intakes and long-term effects of sodium restriction in essential hypertension. Lancet. 1989 Nov 25;2(8674):1244-7. doi: 10.1016/s0140-6736(89)91852-7. PMID 2573761
- [Background] Piovesana Pde M, Sampaio Kde L, Gallani MC. Association between Taste Sensitivity and Self-Reported and Objective Measures of Salt Intake among Hypertensive and Normotensive Individuals. ISRN Nutr. 2012 Oct 24;2013:301213. doi: 10.5402/2013/301213. eCollection 2013. PMID 24967247
- [Background] Kusaba T, Mori Y, Masami O, Hiroko N, Adachi T, Sugishita C, Sonomura K, Kimura T, Kishimoto N, Nakagawa H, Okigaki M, Hatta T, Matsubara H. Sodium restriction improves the gustatory threshold for salty taste in patients with chronic kidney disease. Kidney Int. 2009 Sep;76(6):638-43. doi: 10.1038/ki.2009.214. Epub 2009 Jun 10. PMID 19516246